CLINICAL TRIAL: NCT07362680
Title: Effects of Ultrasound-guided Recruitment Manoeuvres on Postoperative Pulmonary Complications in OSA Patients Undergoing Total Laparoscopic Hysterectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EC-25-117
Record Dates: First submitted 2025-12-18; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Total Laparoscopic Hysterectomy; Atelectasis, Postoperative
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the SRM group (Active Comparator): the sustained inflation recruitment maneuver group, n=30
  Interventions: Procedure: the sustained inflation recruitment maneuver
- the PRM group (Active Comparator): the incremental PEEP recruitment maneuver group, n=30
  Interventions: Procedure: the incremental PEEP recruitment maneuver
- the URM group (Experimental): the Ultrasound-guided recruitment maneuver group, n=30
  Interventions: Procedure: the Ultrasound-guided recruitment maneuver

INTERVENTIONS:
Procedure: the sustained inflation recruitment maneuver — The APL valve on the anaesthesia machine will be adjusted to 30 cmH₂O, and the rapid oxygen inflow valve will be pressed to increase the pressure to the maximum, maintaining the pressure for 30 seconds.
  Arms: the SRM group
Procedure: the incremental PEEP recruitment maneuver — Starting from 5 cmH₂O, PEEP will be titrated upwards in 5 cmH₂O increments every 30 seconds until a maximum of 30 cmH₂O is reached. After maintaining for 40 seconds, PEEP will be decreased by 5 cmH₂O every 30 seconds until it returns to the pre-recruitment level.
  Arms: the PRM group
Procedure: the Ultrasound-guided recruitment maneuver — Lung ultrasound will be performed on patients. If any lung region has an LUS score ≥ 2, ultrasound-guided RM will be performed; otherwise, no operation will be conducted. After the ultrasound examination, the probe will be positioned over the lung region exhibiting the most severe aeration loss (highest LUS) to guide the RMs. The ventilator will be set to pressure-controlled ventilation (PCV), maintaining the inspiratory pressure at 40 cmH₂O. PEEP will be gradually increased from 5 cmH₂O, with increments of 5 cmH₂O every 5-10 seconds, until ultrasound shows no atelectatic areas. The pressure will be maintained at 40 cmH₂O for 40 seconds. An airway pressure ceiling of 40 cmH₂O was established, and the pressure and the time used for the RM will be recorded.
  Arms: the URM group

SUMMARY:
This study aims to evaluate the lung-protective effects of ultrasound-guided lung recruitment maneuvers in patients with OSA undergoing total laparoscopic hysterectomy and to explore the efficacy of EELV measurement in assessing the effectiveness of these maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Scheduled for elective total laparoscopic hysterectomy;
* American Society of Anesthesiologists (ASA) I to III;
* BMI > 28 kg/m²;
* STOP-BANG score ≥ 3.

Exclusion Criteria:

* Abnormal findings on preoperative chest X-ray or CT, such as atelectasis, pneumothorax, thoracic deformity, pleural effusion, or neuromuscular diseases;
* Pre-existing severe pulmonary diseases;
* Severe cardiac arrhythmias or a history of cardiac surgery;
* Allergy to any medications used in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The lung ultrasound scores of patients after endotracheal intubation (T1), after the first lung recruitment procedure (T2), after the operation (T3), after the second lung recruitment procedure (T4), and 30 minutes after extubation (T5) | Perioperative

SECONDARY OUTCOMES:
Recruitment volume measured by the ΔEELV method | Perioperative

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT07362680/Prot_SAP_000.pdf